CLINICAL TRIAL: NCT03398928
Title: Delirium Treatment With Acupuncture in Internal Medicine Departments: a Randomized Sham-controlled Clinical Trial
Brief Title: Delirium Treatment With Acupuncture in Internal Medicine Departments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0102-14-BNZ
Record Dates: First submitted 2017-12-31; First posted 2018-01-16 (Actual); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2017-12

CONDITIONS: Delirium in Old Age
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture for delirium treatment
  Interventions: Other: Acupuncture
- Standard care (No Intervention): Standard conventional delirium care at the discretion of the department medical staff

INTERVENTIONS:
Other: Acupuncture — Acupuncture added to usual care
  Arms: Acupuncture

SUMMARY:
Delirium frequently occurs in hospitalized older people, and treatment options are limited. Acupuncture has been shown to reduce agitation in the setting of dementia. The investigators will test the hypothesis that it may also assist in treating delirium.

DETAILED DESCRIPTION:
This randomized-controlled trial aims to evaluate the efficacy of acupuncture integrated with standard care as compared to standard care only for the treatment of delirium in hospitalized older persons.

Patients aged 65 and older, hospitalized in the internal medicine departments of Bnai Zion Medical Center and diagnosed with delirium or subsyndromal delirium will be randomized to either true acupuncture with usual care, or usual care only. Daily treatments and outcomes' follow-up will be conducted up to one week from recruitment or until resolution of delirium or subsyndromal delirium for 48 hours. The primary outcome will be delirium resolution evaluated as time-to-first delirium remission (over 7 days) and the number of days spent delirium-free.Side effects will be monitored daily.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in internal medicine department
* Aged over 65 years
* Delirium or subsyndromal delirium within the last 48 hours

Exclusion Criteria:

* Platelet count under 20x10^9/L
* Encephalopathy explained by a cause other than delirium (acute stroke, alcohol, cirrhosis, etc.)
* History of severe dementia
* Communication barriers preventing delirium assessment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elad Schiff, M.D., Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Golomb 47, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levy I, Gavrieli S, Hefer T, Attias S, Schiff A, Oliven R, Wisberg-Levi S, Hanchinsky R, Schiff E. Acupuncture Treatment of Delirium in Older Adults Hospitalized in Internal Medicine Departments: An Open-Label Pragmatic Randomized-Controlled Trial. J Geriatr Psychiatry Neurol. 2022 May;35(3):333-343. doi: 10.1177/0891988721996804. Epub 2021 Mar 9. PMID 33685268

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupuncture: Acupuncture for delirium treatment
  Acupuncture + Standard care
Period: Overall Study
Arm/Group | Acupuncture | Standard Care
Started | 50 | 31
Completed | 50 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Standard Care | Total
Number analyzed (Participants) | 50 | 31 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 84 (7.8) | 85.3 (6.7) | 84 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 12 | 37
  Male | 25 | 19 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Long CAM-Severity (minimum: 0, better prognosis; maximum: 19, worse prognosis) [Median (Full Range); unit: units on a scale] | 8 [3 to 15] | 9 [4 to 14] | 8 [3 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Number of Delirium-free Days During the 7 Days of Evaluation
Description: Number of delirium-free days, based on daily assessment of Confusion Assessment Method scale - a validated diagnostic tool addressing the four features of delirium (acute and fluctuating course, inattention, disorganized thinking and impaired level of consciousness). Definite delirium is defined as the first two features plus either one of the third or fourth, while subsyndromal delirium includes patients not meeting these diagnosis criteria but displaying two or more of these four features including the first one (acute and fluctuating course).
Time Frame: At baseline, day 2, day 3, day 4, day 5, day 6 and day 7 of the study
Measure: Median (Full Range); unit: days
Arm/Group | Acupuncture | Standard Care
Number analyzed (Participants) | 50 | 31
days | 5.5 [0 to 6] | 0 [0 to 6]
Statistical Analysis 1: Comparison: Acupuncture vs Standard Care; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Time-to-first Remission of Delirium in the 7 Days of Evaluation
Description: Daily assessment of Confusion Assessment Method scale - a validated diagnostic tool addressing the four features of delirium (acute and fluctuating course, inattention, disorganized thinking and impaired level of consciousness). Definite delirium is defined as the first two features plus either one of the third or fourth, while subsyndromal delirium includes patients not meeting these diagnosis criteria but displaying two or more of these four features including the first one (acute and fluctuating course).
Time Frame: At baseline, day 1, day 2, day 3, day 4, day 5, day 6, day 7 of the study
Measure: Median (Full Range); unit: days
Arm/Group | Acupuncture | Standard Care
Number analyzed (Participants) | 50 | 31
days | 1 [1 to 7] | 7 [1 to 7]
Statistical Analysis 1: Comparison: Acupuncture vs Standard Care; Test type: Superiority; p < 0.001, Log Rank

3. Secondary Outcome: Length of Hospital Stay
Description: Days of hospitalization
Time Frame: Through study completion, an average of 2-3 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Acupuncture | Standard Care
Number analyzed (Participants) | 50 | 31
days | 16.4 (14.7) | 18.3 (15)

4. Secondary Outcome: Functional Status at Discharge
Description: Total Katz Activity of Daily Living (ADL) score at discharge - score assessing activities of daily living, minimum: 0 (worse prognosis), maximum: 6 (best prognosis), calculated as the sum of the following activities (1: independence, 0: dependence): bathing, dressing, toileting, transferring, continence, feeding.
Time Frame: Through study completion, an average of 2-3 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Acupuncture | Standard Care
Number analyzed (Participants) | 50 | 31
units on a scale | 2 [0 to 6] | 3.5 [0 to 6]

5. Secondary Outcome: Delirium Severity
Description: Comparison of the sum of long Confusion Assessment Method (CAM-S) score from day 2 (before treatment in the second day of the study) until day 7 (last day of evaluation). CAM-S scale includes 10 delirium-related items, the first one being rated on a 0-1 scale and the nine followings in a 0-2 scale for a total 0-19 score. Higher scores indicate worse outcomes. When summed across 7 days, the total scale range is 0-133 with 0-3 being no delirium, 4-6 being low severity, 7-13 being moderate severity and +/=14 being high severity (Vasunilashorn SM, Marcantonio ER, Gou Y, et al. Quantifying the Severity of a Delirium Episode Throughout Hospitalization: the Combined Importance of Intensity and Duration. J Gen Intern Med. 2016;31(10):1164-1171).
Time Frame: Sum of CAM-S at day 2 + day 3 + day 4 + day 5 + day 6 + day 7 of the study
Population: Long CAM-S sum was missing for some participants (5 in the acupuncture arm, and 3 in the standard care arm)
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard Care
Number analyzed (Participants) | 45 | 28
Participants
  No delirium (Long CAM-S sum = 0-3) | 11 | 3
  Low severity (Long CAM-S sum = 4-6) | 6 | 0
  Moderate severity (Long CAM-S sum = 7-13) | 9 | 1
  High severity (Long CAM-S sum >= 14) | 19 | 24
Statistical Analysis 1: Comparison: Acupuncture vs Standard Care; Test type: Superiority; p = 0.002, Chi-squared — The statistical analysis applies to all the rows

6. Secondary Outcome: Number of Days in Which Antipsychotic Drugs Were Used
Description: Daily patient chart review for antipsychotic drugs
Time Frame: At baseline, day 2, day 3, day 4, day 5, day 6 and day 7 of the study
Measure: Median (Full Range); unit: days
Arm/Group | Acupuncture | Standard Care
Number analyzed (Participants) | 50 | 31
days | 7 [0 to 7] | 7 [0 to 7]
Statistical Analysis 1: Comparison: Acupuncture vs Standard Care; Test type: Superiority; p = 0.253, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Visual Assessment Scale (VAS) for Pain
Description: Daily Visual Assesment Scale - This scale measures pain in a 0-10 score. Higher scores indicate worse pain.
Time Frame: At baseline, day 2, day 3, day 4, day 5, day 6 and day 7 of the study
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Acupuncture | Standard Care
Number analyzed (Participants) | 50 | 31
units on a scale
  Day 1 | 0 [0 to 10] | 0 [0 to 5]
  Day 2 | 0 [0 to 2] | 0 [0 to 0]
  Day 3 | 0 [0 to 5] | 0 [0 to 5]
  Day 4 | 0 [0 to 6] | 0 [0 to 3]
  Day 5 | 0 [0 to 6] | 0 [0 to 4]
  Day 6 | 0 [0 to 10] | 0 [0 to 5]
  Day 7 | 0 [0 to 10] | 0 [0 to 0]

8. Secondary Outcome: Sleep
Description: Confusion Assessment Method Severity (CAM-S) scale, tenth item: "sleep-wake cycle". The CAM-S includes 10 delirium-related items, the first one being rated on a 0-1 scale and the nine followings in a 0-2 scale for a total 0-19 score. Here we will use the tenth item (sleep-wake cycle) rated on a 0-2 scale, higher scores indicating worse outcomes.
Time Frame: At baseline, day 2, day 3, day 4, day 5, day 6 and day 7 of the study
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Acupuncture | Standard Care
Number analyzed (Participants) | 50 | 31
units on a scale
  Day 1 | 1 [0 to 2] | 1 [0 to 2]
  Day 2 | 0 [0 to 2] | 1 [0 to 2]
  Day 3 | 0 [0 to 2] | 0 [0 to 2]
  Day 4 | 0 [0 to 2] | 0 [0 to 0]
  Day 5 | 0 [0 to 1] | 0 [0 to 2]
  Day 6 | 0 [0 to 0] | 0 [0 to 2]
  Day 7 | 0 [0 to 0] | 0 [0 to 2]

9. Secondary Outcome: Delirium Complications
Description: Falls, pulling out lines, pressure ulcers, physical restraints
Time Frame: At baseline, day 2, day 3, day 4, day 5, day 6 and day 7 of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard Care
Number analyzed (Participants) | 50 | 31
Participants
  Fall | 1 | 1
  Need for physical restraints due to agitation | 5 | 5
  Pulling-out IV lines | 3 | 2
  Pulling-out urinary catheter | 1 | 1
  Pressure ulcers worsening | 1 | 1

10. Secondary Outcome: Mortality
Description: Patient death
Time Frame: During the 7-day intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Standard Care
Number analyzed (Participants) | 50 | 31
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Acupuncture | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/31
Other Adverse Events (participants affected / at risk) | 9/50 | 7/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acupuncture (N=50) | Standard Care (N=31)
Fall (Injury, poisoning and procedural complications) | 1 | 1
Pulling-out IV lines (Injury, poisoning and procedural complications) | 3 | 2
Pulling-out urinary catheter (Injury, poisoning and procedural complications) | 1 | 1
Pressure ulcers worsening (Skin and subcutaneous tissue disorders) | 1 | 1
Need for physical restraints due to extreme agitation (Injury, poisoning and procedural complications) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT03398928/Prot_SAP_000.pdf